CLINICAL TRIAL: NCT06667258
Title: Hearables: Ear Electrocardiography (ECG) and Photoplethysmography (PPG) for Real-time Detection of Cardiac Arrhythmias
Brief Title: Hearables: Ear-ECG and PPG for Detection of Cardiac Arrhythmias
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 22HH7866; 318229 (Other: IRAS)
Record Dates: First submitted 2024-10-24; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy: Volunteers who have not been diagnosed with any heart rhythm problems, or patients whose heart rhythm issues are not showing up at the time of recruitment.
  Interventions: Device: Ear ECG/PPG sensors
- Arrhythmia patients: Patients who have been previously diagnosed with an abnormal heart rhythm and are showing signs of it when they join the study.
  Interventions: Device: Ear ECG/PPG sensors

INTERVENTIONS:
Device: Ear ECG/PPG sensors — Medical graded electrodes placed in the mastoid, in-ear foam-based earpiece (like commercial earplugs) with cloth electrodes, off-the-shelf pulse oximeter placed behind the ear

SUMMARY:
The goal of this observational study is to determine the feasibility of detecting abnormal heart rhythms, known as arrhythmias, by recording Electrocardiogram (ECG) and Photoplethysmogram (PPG) waveforms from the ears in patients who have already been diagnosed with arrhythmias. The main questions it aims to answer are:

* Can ECG and PPG signals from the ears reliably detect arrhythmias?
* How do ear-based ECG/PPG waveforms compare to standard single-lead ECG in detecting abnormal rhythms?

Researchers will compare data from healthy controls and arrhythmia patients to see if ear-based recordings are as effective as traditional methods.

DETAILED DESCRIPTION:
The main goal of this study is to determine the feasibility of detecting abnormal heart rhythms, known as arrhythmias, by recording Electrocardiogram (ECG) and Photoplethysmogram (PPG) waveforms from the ears.

The study includes both healthy control subjects and patients who have already been diagnosed with arrhythmias. These individuals will be approached by a clinical member of the research team during their hospital stay or outpatient visit at Imperial College NHS Trust (ICHNT). Patients will be given comprehensive information about the study through a patient information sheet and will be asked for their written informed consent, with adequate time provided for questions and understanding.

To capture Ear-ECG/PPG waveforms, a variety of standard medical-grade sensors and electrodes will be placed in and around both ears. These include standard EEG electrodes on each mastoid secured with medical-grade gel, and an in-ear foam-based earpiece (like commercial earplugs) with cloth electrodes. An additional PPG sensor (MAX30101 from Maxim Integrated) will be attached to the back of the ear with adhesive medical tape. The patient will also be connected to a standard single-lead ECG and a blood pressure cuff, already part of their standard care on the hospital ward.

Once the setup is complete, each patient will follow 3 different recording protocols displayed on a screen. Patients will be asked to sit upright (Protocol 1) and engage in a series of simple activities with designated breaks in between, including head movements, counting aloud to 60, chewing gum (or simulating chewing), walking (if able) freely under medical supervision with assistance if needed (Protocol 2), slow controlled breathing and immersing their hand in cold water (Protocol 3). The total recording time including setup will be approximately 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent;
* Healthy and diagnosed with cardiac arrhythmias.

Exclusion Criteria:

* No abnormal ear anatomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 healthy patients and 50 patients with an established diagnosis of cardiac arrhythmias
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of arrhythmia detection in the group of participants | Up to 6 months from study completion
  Accuracy in detecting and classifying arrhythmias from signals recorded from the ears of patients with or without arrhythmia (Protocol 1)

SECONDARY OUTCOMES:
Signal to Noise Ratio | Up to 6 months from study completion
  The Signal quality of Ear-ECG expressed as Signal to Noise ratio evaluated against 1-lead 'Rhythm strip' ECG at rest (Protocol 1)
Signal quality improvement after artefact removal (expressed as difference) | Up to 6 months from study completion
  Noise reduction from Ear-ECG and Ear-PPG after removal of artefacts that may be due to movement (Protocol 2)
Error in blood pressure estimation by comparing ear-ECG and ear-PPG signals | Up to 6 months from study completion
  Accuracy of estimating blood pressure by subtracting the ear-ECG and ear-PPG peak time location (Protocol 3)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas S. Peters, MD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, Non-US/Non-Canadian, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Held within Imperial College London as per standard local data protection guidelines. Data may be considered for sharing upon reasonable request.

REFERENCES:
- [Background] von Rosenberg W, Chanwimalueang T, Goverdovsky V, Peters NS, Papavassiliou C, Mandic DP. Hearables: feasibility of recording cardiac rhythms from head and in-ear locations. R Soc Open Sci. 2017 Nov 15;4(11):171214. doi: 10.1098/rsos.171214. eCollection 2017 Nov. PMID 29291107

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-30): https://cdn.clinicaltrials.gov/large-docs/58/NCT06667258/Prot_SAP_000.pdf